CLINICAL TRIAL: NCT07147426
Title: A Prospective, Randomized Controlled, Phase II Clinical Study on the Neoadjuvant Treatment of Locally Advanced Resectable Head and Neck Squamous Cell Carcinoma With Tislelizumab Combined With Chemotherapy for Different Cycles (NeoTempo)
Brief Title: Tislelizumab Combined With Chemotherapy for Different Cycles of Neoadjuvant Therapy for Locally Advanced Resectable Squamous Cell Carcinoma of the Head and Neck (NeoTempo)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Xudong Wang, Tianjin Medical University Cancer Institute and Hospital, Tianjin Medical University Cancer Institute and Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20250855
Record Dates: First submitted 2025-08-20; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Head &Amp; Neck Squamous Cell Carcinoma
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 cycles arm (Experimental)
  Interventions: Drug: Tislelizumab Combined With Chemotherapy for 4 cycles
- 2 cycles arm (Active Comparator)
  Interventions: Drug: Tislelizumab Combined With Chemotherapy for 2 cycles

INTERVENTIONS:
Drug: Tislelizumab Combined With Chemotherapy for 4 cycles — Tislelizumab: 200mg, day 1, every 3 weeks for 4 cycles Cisplatin: 75mg/m^2 Nab-paclitaxel: 260mg/m^2
  Arms: 4 cycles arm
Drug: Tislelizumab Combined With Chemotherapy for 2 cycles — Tislelizumab: 200mg, day 1, every 3 weeks for 2 cycles Cisplatin: 75mg/m^2 Nab-paclitaxel: 260mg/m^2
  Arms: 2 cycles arm

SUMMARY:
This study aims to explore the optimal course of neoadjuvant immunotherapy for HNSCC by comparing the efficacy and safety of 4 cycles and 2 cycles of neoadjuvant tislelizumab combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or pathological diagnosis of head and neck squamous cell carcinoma;
* Initially resectable stage III-IVB oral cancer/laryngeal cancer/hypopharyngeal cancer/P16-oropharyngeal cancer, or stage III p16+ oropharyngeal cancer (AJCC 8th), and evaluated by the researcher to achieve R0 resection;
* Plan to perform neoadjuvant therapy;
* No previous anti-tumor treatment for HNSCC;
* There is at least one measurable lesion;
* Eastern Cooperative Oncology Group Performance Status (ECOG) score 0-2;
* The expected survival period is ≥3 months
* The functions of vital organs meet the following requirements (excluding any blood components and cell growth factors used within 7 days) :

  i. Normal bone marrow reserve function, white blood cell (WBC) ≥3.0×109/L; Neutrophil count (NEUT) ≥ 1.5×109/L, platelet count (PLT) ≥100×109/L, hemoglobin (Hb) ≥90 g/L; ii. Normal renal function or serum creatinine (SCr) ≤ 1.5 times the upper limit of normal value (ULN) or creatinine clearance rate ≥50 ml/min (Cockcroft-Gault formula); iii. Normal liver function or total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); The level of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is ≤ 2.5 times the upper limit of the normal value (ULN).
* Be able to and willing to abide by the research and follow-up procedures;
* Men and women of gestational age must agree to take adequate contraceptive measures throughout the study period and within 6 months after the end of treatment.
* The patient voluntarily joined this clinical study, signed the informed consent form, had good compliance and was able to cooperate with the follow-up.

Exclusion Criteria:

* Previously received anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on T-cell co-stimulation or checkpoint pathways);
* There is a clear history of allergies, and there may be potential allergies or intolerances to the research drug and its similar biological agents;
* Participated in clinical trials of other anti-tumor drugs within 4 weeks before the first administration; Or within 4 weeks before the first administration or planning to receive a live attenuated vaccine during the study period;
* Other malignant tumors have occurred within the past five years (except for well-treated squamous cell carcinoma of the skin or controlled basal cell carcinoma of the skin);
* Immunosuppressive drugs have been used within 14 days prior to the first use of tislelizumab, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroid hormones (i.e., no more than 10 mg/ day of prednisolone or equivalent physiological doses of other corticosteroids).
* Advanced patients with symptoms, who have spread to internal organs and are at risk of life-threatening complications in the short term (including those with uncontrollable large amounts of exudate [thoracic, pericardial, abdominal], pulmonary lymphangitis and more than 30% liver involvement)
* Any active autoimmune diseases or a history of autoimmune diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or those whose asthma has completely relieved in childhood and do not require any intervention in adulthood can be included; Asthma subjects who require bronchodilators for medical intervention cannot be included.
* Suffering from grade II or above myocardial ischemia or myocardial infarction, and poorly controlled arrhythmias (including QTc interval ≥450ms in men and ≥470ms in women). According to the NYHA standard, patients with grade Ⅲ to Ⅳ cardiac failure, or those whose left ventricular ejection fraction (LVEF) is less than 50% as indicated by echocardiography; Myocardial infarction occurred within 6 months before enrollment, New York Heart Association Class II or above heart failure, uncontrolled angina pectoris, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease, or electrocardiogram indicating acute ischemia or abnormal active conduction system
* Concurrent severe infection within 4 weeks before the first administration (e.g., requiring intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever >38.5°C during the screening period/before the first administration;
* Those with a history of abuse of psychotropic drugs and unable to quit, or those with mental disorders;
* Major surgical operations have been performed within 4 weeks prior to the first administration. Or have an open wound or fracture;
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (positive hepatitis C antibody and HCV-RNA higher than the detection limit of the analytical method), or co-infection with hepatitis B and hepatitis C;
* There is central nervous system metastasis;
* Those with a history of hereditary or acquired bleeding or coagulation disorders (the specific inclusion is determined by the researcher);
* Other circumstances where the researcher determines that one is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | 6 months
  Pathological complete response (pCR) is defined as having no residual invasive squamous cell carcinoma within the resected primary tumor specimen.

SECONDARY OUTCOMES:
Major Pathological Response (mPR) | 6 months
  The percentage of participants with a major pathological response (mPR) is defined as ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen.
Organ perservation rate | 6 months
  Organ perservation rate defined as the proportion of patients who successfully preserved their organs and functions through neoadjuvant treatment.
Operation delay rate | 6 months
  Operation delay rate defined as any change to scheduled surgery date considered to be at least possibly related to neoadjuvant treatment.
Objective resopnse rate (ORR) | 6 months
  ORR defined as the proportion of all subjects who achieved complete response (CR) or partial response (PR) as assessed by RECIST V1.1 after the end of neoadjuvant therapy
Event-free Survival (EFS) | 3 years
  EFS is the time from the date of randomization to the date of first record of any of the following events: radiographic disease progression; local or distant progression or recurrence as assessed with imaging or biopsy as indicated; or death due to any cause.
Overall Survival (OS) | 3 years
  OS is the time from randomization to death due to any cause.
Percentage of adverse events graded by CTCAE v5.0 | 3 years
  Percentage of adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).
Change From Baseline in Quality of Life Scale (QoL) (EORTC QLQ-C30) items 30 | 3 years
  Change from baseline in the combined score of quality of life (QoL) using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (EORTC QLQ-C30) items 30
Change From Baseline in Quality of Life Scale (QoL) EOTRC QLQ -H&N 35 | 3 years
  Change from baseline in the combined score of quality of life (QoL) using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire EOTRC QLQ -H&N 35

IPD SHARING:
Plan to Share IPD: No